CLINICAL TRIAL: NCT05962086
Title: Determining Developmental and Clinical Markers Affecting Urinary Function of Children With Spinal Dysraphism: A Multicenter, Retrospective Cohort
Brief Title: Determining Developmental and Clinical Markers Affecting Urinary Function of Children With Spinal Dysraphism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Severance Hospital (Other); Samsung Medical Center (Other); Keimyung University Dongsan Medical Center (Other); Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kwanjin Park, Professor, Seoul National University Hospital
Other Study IDs: 2210-092-1369
Record Dates: First submitted 2023-06-10; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Spinal Dysraphism
Keywords: Spina Bifida; Neurogenic Bladder; Neurogenic Detrusor Overactivity; Detrusor Overactivity; Incontinence
MeSH Terms: conditions — Spinal Dysraphism; Urinary Bladder, Neurogenic; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify developmental and clinical biomarkers that affect urinary incontinence at the ages of 5, 7, and 10 according to different neuro-urological clinical factors.

DETAILED DESCRIPTION:
This retrospective observational cohort study aims to identify developmental and clinical biomarkers that affect urinary incontinence at the ages of 5, 7, and 10 according to the types of spinal dysraphism, conus medullaris location, and urodynamics test results.

ELIGIBILITY:
Inclusion Criteria:

- Those who received spinal dysraphism diagnosis (ICD Code: Q05.1-05.9) and have been following up and receiving treatments due to neurogenic bladder.

Exclusion Criteria:

- As the study is a retrospective study, there is no exclusion criteria.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Spinal dysraphism (SD) is a congenital abnormality that results in an abnormal structure in the spine, including the bony structure, the spinal cord, and the nerve roots. Patients with SD often suffer from multiple complications such as neurological problems, urological problems, orthopedic problems, and pain. A numerous studies have demonstrated that at least 70-90% of the patients experience neurogenic bladder or neurogenic detrusor overactivity, which affects both physical and psychosocial aspects of quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Achieving full continence at age 5 | Age 5
  Achieving full urinary and fecal continence at age 5
Achieving full continence at age 7 | Age 7
  Achieving full urinary and fecal continence at age 7.
Achieving full continence at age 10 | Age 10
  Achieving full urinary and fecal continence at age 10

CONTACTS AND LOCATIONS:
Overall Officials: Kwanjin Park, MD/PHD, Study Chair — Seoul National University Hospital; Sang Woon Kim, MD/PHD, Principal Investigator — Severance Hospital; Sang Hoon Song, MD/PHD, Principal Investigator — Asan Medical Center; Minki Baek, MD/PHD, Principal Investigator — Samsung Medical Center; Jae Min Chung, MD/PHD, Principal Investigator — Pusan National University Yangsan Hospital; Ji Yong Ha, MD/PHD, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (6):
- South Korea (6):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
Not willing to share individual participant data (IPD) for this particular study.